CLINICAL TRIAL: NCT04582318
Title: A Randomized, Double Blind, Placebo Controlled, Combined Phase 1/2 Single Dose and Multiple Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of NGM621 in Healthy Volunteers and the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy in Subjects With Confirmed SARS-CoV-2 Infection
Brief Title: A Phase 1/2 Study to Assess the Safety, Tolerability and Pharmacokinetics of NGM621 in Healthy Subjects, and to Assess the Safety, PK and Efficacy in Subjects With Moderate to Severe ARDS Caused by COVID-19
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the rapidly changing therapeutic landscape in the COVID-19 space and an assessment of unmet medical need, Part 2 of the study was cancelled (per protocol Section 4.3). Meanwhile, Part 1 of the study was completed.
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 621-CP-102
Record Dates: First submitted 2020-10-07; First posted 2020-10-09 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part 1 Dose Level 1 - Active (Experimental)
  Interventions: Biological: NGM621
- Part 1 Dose Level 1 - Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- Part 1 Dose Level 2 - Active (Experimental)
  Interventions: Biological: NGM621
- Part 1 Dose Level 2 - Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- Part 2 Multi-Dose Level 1 - Active (Active Comparator)
  Interventions: Biological: NGM621
- Part 2 Multi-Dose Level 1 - Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- Part 2 Multi-Dose Level 2 - Active (Active Comparator)
  Interventions: Biological: NGM621
- Part 2 Multi-Dose Level 2 - Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NGM621 — NGM621 will be administered via IV infusion
  Arms: Part 1 Dose Level 1 - Active; Part 1 Dose Level 2 - Active; Part 2 Multi-Dose Level 1 - Active; Part 2 Multi-Dose Level 2 - Active
Biological: Placebo — Placebo will be administered via IV infusion
  Arms: Part 1 Dose Level 1 - Placebo; Part 1 Dose Level 2 - Placebo; Part 2 Multi-Dose Level 1 - Placebo; Part 2 Multi-Dose Level 2 - Placebo

SUMMARY:
This study is a combined Phase 1 and Phase 2 study with IV infusion of NGM621 to evaluate the safety, tolerability, and PK in healthy volunteers (Part 1), and safety, tolerability, PK and efficacy in subjects with confirmed SARS-CoV-2 infection (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of childbearing potential must have a negative serum pregnancy test result at Screening and a negative urine pregnancy test result prior to dosing.
* Female subjects of childbearing potential and male subjects with a female partner of childbearing potential must use an effective method of contraception during the study, for at least 1 month following study completion, and must not plan to become pregnant for at least 1 month after her last study medication dose.
* BMI 18-32 kg/m2 inclusive
* Ability to understand and provide informed consent
* Subjects confirmed with SARS-CoV-2 infection by PCR and hospitalized
* If on mechanical support, less or equal than 2 days on mechanical ventilation or oxygenation

Exclusion Criteria:

* Currently enrolled in another investigational protocol to treat SARS-CoV-2 infection
* Known history of complement deficiency
* Active infection with, or history of, compllicated pneumococcal or Neisseria meningitis infection or history of unexplained, recurrent infection, within the last 60 days prior to dosing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events - Part 1 | 85 days
  TEAEs in subjects receiving NGM621 compared to placebo
Treatment emergent adverse events - Part 2 | 91 days
  TEAEs in subjects receiving NGM621 compared to placebo
Clinical status at Day 15 and Day 29 - Part 2 | 29 days
  Clnical status (on an 8-point ordinal scale) in NGM621 group versus placebo group

SECONDARY OUTCOMES:
Maxiumum Serum Concentration [Cmax] | 91 days
Mortality at Day 29 | 29 days
Duration of Supplemental Oxygen Requirement | 91 days
Change in Hemolytic Assays (CH50 and AH50) from Baseline | 91 days

CONTACTS AND LOCATIONS:
Locations (1):
- NGM Clinical Study Site, Brisbane, Australia

IPD SHARING:
Plan to Share IPD: Undecided
This is a proof-of-concept study assessing the safety, tolerability, PK, and efficacy of systemic use of NGM621 versus placebo in both healthy subjects and subjects confirmed with SARS-CoV-2 infection. We will continue to evaluate whether IPD will be shared with other researchers.